CLINICAL TRIAL: NCT01085552
Title: A Phase I Single Centre Open Label Trial to Investigate the Bioequivalence of a Single Subcutaneous Dose of Epoetin Beta (NeoRecormon®) in Healthy Japanese and Caucasian Male Subjects
Brief Title: Bioequivalence of a Single Subcutaneous Dose of Epoetin Beta in Healthy Japanese and Caucasian Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: InCROM Europe Clinical Research (Industry)
Responsible Party: Dr Daryl Bendel, InCROM Europe Clinical Research
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: EICE07060
Record Dates: First submitted 2010-03-11; First posted 2010-03-12 (Estimated); Last update posted 2010-03-12 (Estimated); Status verified 2010-03

CONDITIONS: Chronic Kidney Failure; Anaemia
Keywords: NeoRecormon®; Caucasian; Japanese; Bioequivalence; Ethnic
MeSH Terms: conditions — Kidney Failure, Chronic; Anemia | interventions — epoetin beta

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Other): Group A consists of 11 Caucasian male subjects Group B consists of 12 Japanese male subjects
  Interventions: Drug: Epoetin Beta

INTERVENTIONS:
Drug: Epoetin Beta — Epoetin Beta. A single subcutaneous dose of 50IU/kg on Day 1. The body weight recording on day -1 will be used to calculate the dosage

SUMMARY:
A study to see how a single subcutaneous dose of Epoetin beta (NeoRecormon®) in healthy Japanese compares with a single subcutaneous dose of Epoetin beta (NeoRecormon®) in Caucasian Male subjects. Each subject received a single subcutaneous dose of 50IU/kg of NeoRecormon Multidose solution on Day 1.

DETAILED DESCRIPTION:
Ethnic comparison studies are becoming common research requirements in order to identify differences in response to drugs in various ethnic populations. This study will investigate the pharmacokinetic parameters and pharmacodynamic response in healthy Caucasian and Japanese male subjects after a single subcutaneous administration of 50IU/kg Epoetin beta

This is a Phase I single centre, open label trial to investigate the bioequivalence of a single subcutaneous dose of Epoetin beta (NeoRecormon®) in healthy Japanese and Caucasian Male subjects.

The primary objectives are 1) to establish the pharmacokinetic parameters of Epoetin beta in healthy Japanese and Caucasian males, and 2) to compare the pharmacokinetic parameters AUCinf and Cmax in healthy Japanese and Caucasian males. The secondary objective is to establish the pharmacodynamic parameters of a single dose of Epoetin beta in healthy Japanese and Caucasian males.

Subjects will receive a single subcutaneous administration of 50IU/kg on one occasion only. The planned study duration is approximately 1 month.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male Japanese volunteers (both parents and all four grandparents must be Japanese, and subject must have been born in Japan, subjects should usually reside in Japan but can have been resident outside of Japan for up to 5 years), or Healthy male Caucasian volunteers.
* Aged between 20 and 40 years of age.
* Body weight of 50kg - 80 kg inclusive with a Body mass index (BMI) between 18 - 29 kg/m2 inclusive at screening.
* Subjects must be in good health as determined by a medical history, medical examination, electrocardiogram, serum biochemistry, haematology, serology and urinalysis.
* Provide their written informed consent to participate in the trial after reading the information and consent form, and after having opportunity to discuss the trial with the investigator or delegate.
* Sufficient intelligence to understand the nature of the trial and any hazards of participating in it. Ability to communicate satisfactorily with the investigator and/or delegate and participate in, and comply with the requirement's of the entire trial.
* Willing to abstain from Alcohol consumption from 48 hours before trial drug administration until last outpatient visit.
* Subjects must be willing to use one of the following methods of contraception from the first dose of trial medication until completion of follow-up procedures:In addition to the use of condom and spermicide (foam/gel/film), male subjects without a vasectomy must assure that their female partner uses another form of contraception such as an IUD, diaphragm or hormonal contraception if the female partner could become pregnant from the time of the first dose of trial medication until one month after the follow up visit.
* Have an upper limit of14g/dL for haemoglobin, 45% for Hematocrit and 1.9% for Reticulocytes.
* Have normal safety results for Creatinine, Liver function tests, serum Ferritin, Folic acid and vitamin B12 at the screening assessment

Exclusion Criteria:

* Clinically relevant abnormal history, physical findings, ECG, or laboratory values at the screening visit that could interfere with the objective of the trial or the safety of the volunteer.
* Clinically significant illness within 4 weeks prior to the screening visit.
* Subjects with past or present histories of liver disease, angina, renal disease, hypertension, epilepsy, cardiovascular, cerebrovascular, thrombocytosis or peripheral vascular disease.
* Subjects who have used any systemic, topical prescription, non-prescription or herbal medication within 14 days of start of dosing with the exception of paracetamol up to 3g per day.
* Subjects who smoke more than 5 cigarettes per day.
* Subjects who have donated 400ml of blood during the 1 month before dosing.
* Subjects who have received an investigational product 3 months preceding the trial.
* Subjects who have a clinically significant history of drug hypersensitivity or allergic disease.
* Subjects who consume more than 28 units of alcohol per week or who have history of alcoholism or evidence of drug/chemical abuse. (one unit of alcohol equals ½ pint [285 ml] of beer or lager, one glass [125 ml] of wine or l [25ml] of spirits)
* Subjects who consume excessive amounts of caffeine (more than 5 cups or equivalent per day.
* Subjects with a positive urine drug screen at the screening visit or admission.
* Subjects with known history or evidence of hepatitis B, hepatitis C or HIV1 or HIV2.
* Subjects who in the opinion of their GP or the investigator should not participate in the study.
* Possibility that the subject will not cooperate with the requirements of the protocol as set out in the volunteer information.
* Subjects with any previous exposure to erythropoietin

Ages: 20 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2007-11; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
To establish the pharmacokinetic parameters of Epoetin beta in healthy Japanese and Caucasian males. | 21 Oct 2008
To compare the pharmacokinetic parameters AUCinf and Cmax in healthy Japanese and Caucasian males. | 21 Oct 2008

SECONDARY OUTCOMES:
To establish the pharmacodynamic parameters of a single dose of Epoetin beta in healthy Japanese and Caucasian males. | 21 Oct 2008

CONTACTS AND LOCATIONS:
Overall Officials: Daryl Bendel, MBChB MBA, Principal Investigator — InCROM Clinical Research Unit